CLINICAL TRIAL: NCT06307977
Title: Couples Motivational Interviewing to Reduce Drug Use and HIV Risk in Vulnerable Male Couples
Acronym: CHP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA059272 (NIH)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Substance Use; HIV Infections
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized controlled trial design to evaluate the efficacy of couples motivational interviewing (MI) to reduce the frequency and severity of illicit drug use and frequency of HIV transmission risk behavior (TRB). Participants are randomized to one of two conditions: couples MI or standard couples HIV testing and counseling (CHTC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention: CHTC as usual (No Intervention): Participants complete the standard Couples HIV Testing and Counseling session (CHTC).
- Behavioral: Couples Health Project (Active Comparator): A three-session intervention for couples addressing couples communication skills, substance use, sexual agreements. The intervention also includes couples HIV testing and counseling in the final session.
  Interventions: Behavioral: Couples Health Project

INTERVENTIONS:
Behavioral: Couples Health Project — A 3-session, couples motivational Interviewing drug use and HIV risk reduction intervention
  Other Names: CHP
  Arms: Behavioral: Couples Health Project

SUMMARY:
This study utilizes a randomized controlled trial design to evaluate the efficacy of couples motivational interviewing (MI) to reduce the frequency and severity of illicit drug use and frequency of HIV transmission risk behavior (TRB). Participants are randomized to one of two conditions: couples MI or standard couples HIV testing and counseling (CHTC).

ELIGIBILITY:
Inclusion Criteria:

* Have a main partner who is another cisgender male and have been in a relationship for 3 month or longer
* Index participant must be between 18 and 55; Main partner can be any age 18 and older
* One participant must be HIV negative (as confirmed by rapid test)
* One participant must have used at least 1 drug in the past 30 days (cocaine/crack, opiates, misuse of prescription medication, stimulants, psychedelics, ecstasy, ketamine, GHB, amyl nitrite)
* Index participant must have engaged in TRB in the past 30 days- Defined as CAS with a casual partner, or a serodiscordant or non-monogamous main partner
* Live in the United States
* Speak and read English

Exclusion Criteria

* Any signs of serious mental illness or cognitive deficit
* Current suicidal/homicidal ideations
* History of IPV with their main partner and safety concerns in the current relationship.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both partners in the couple must identify as male.
Enrollment: 360 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Drug use Frequency | 9 Months
  Number of reported days of illicit drug use (amphetamines, cocaine/crack, GHB, ketamine or ecstasy) reported on quarterly timeline follow-back assessments
Urine assay for drug use | 9 Months
  Positive urine screen for drug use assessed bi-annually
CAS with casual partners | 9 Months
  Number of total anal sex acts (insertive and receptive) with casual partners reported on quarterly timeline follow-back assessments in the absence of adequate PrEP coverage

SECONDARY OUTCOMES:
Bacterial sexually transmitted infections | 9 Months
  Any chlamydia or gonorrhea diagnosis
Binge Drinking | 9 Months
  Number of days on which 5 or more drinks containing alcohol were reported on the quarterly timeline follow-back interview
PrEP Uptake | 9 months
  self-reported receipt of a PrEP-prescription

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Wayne State University, Detroit, Michigan
  - Hunter College, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Starks TJ, Hillesheim JR, Castiblanco J, Robles G, S Ingersoll K, Outlaw AY, Cain D. A protocol for a randomized controlled trial of couples motivational interviewing to reduce drug use and HIV transmission risk among male couples in the US: the Couples Health Project. BMC Public Health. 2024 Nov 19;24(1):3216. doi: 10.1186/s12889-024-20719-y. PMID 39563247